CLINICAL TRIAL: NCT02894866
Title: Effect of Hyperbaric Oxygen Therapy on Neonatal Hypoxic-Ischemic Encephalopathy
Brief Title: Hyperbaric Oxygen Therapy Improves Outcome of Hypoxic-Ischemic Encephalopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFEC-2016-097
Record Dates: First submitted 2016-08-26; First posted 2016-09-09 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Hypoxic-ischemic Encephalopathy
Keywords: hypoxic-ischemic encephalopathy; hyperbaric oxygen therapy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hyperbaric oxygen (Experimental): Newborns with hypoxic ischemic encephalopathy treated with intensive care and hyperbaric oxygen
  Interventions: Device: hyperbaric oxygen
- control (No Intervention): Newborns with hypoxic ischemic encephalopathy treated with intensive care only

INTERVENTIONS:
Device: hyperbaric oxygen — The hyperbaric oxygen treatment will be administered for 60 min in a baby hyperbaric oxygen chamber pressured with 100% oxygen to 1.5 to 1.8 atm absolute (ATA) and a constant oxygen flow was given to maintain the oxygen. concentration in the chamber at 80% or greater.The treatment will be administered once a day within 7 days after birth, 7 days is a course of treatment, at least for 4 courses.
  Arms: hyperbaric oxygen

SUMMARY:
The purpose of this study is to to evaluate the safety and efficacy of hyperbaric oxygen in term gestation newborn infants with hypoxic-ischemic encephalopathy..

DETAILED DESCRIPTION:
Hypoxic-ischemic encephalopathy (HIE) remains a major cause of neonatal death and long term disabilities. Data from animal studies have shown protective effects of hyperbaric oxygen therapy to impaired brain. Recently research priorities have moved from bench to bedside. Several studies have shown a trend for brain protection of hyperbaric oxygen therapy has emerged as a promising treatment for HIE. Therefore,the investigators organized a multi-centered randomized controlled trial of hyperbaric oxygen therapy in HIE newborn infants.

ELIGIBILITY:
* Inclusion Criteria:

  * Newborn infants whose gestational age ≥37 weeks' gestation, weighing over 2500 g ;
  * Acute perinatal event (e.g., late or variable decelerations, cord prolapse, cord rupture, uterine rupture, maternal trauma, hemorrhage, or cardiorespiratory arrest)
  * With an Apgar score ≤ 3 at one minute and ≤5 at five minutes, and/or a potential of hydrogen of 7.0 or less or a base deficit of 16 mmol per liter or more in a sample of umbilical-cord blood or any blood during the first hour after birth.
  * Having moderate-to-severe encephalopathy (indicated by lethargy, stupor, or coma) and either hypotonia, abnormal reflexes (including oculomotor or pupillary abnormalities), an absent or weak suck, or clinical seizures, and/or have abnormal background activity of at least 20 minutes' duration or seizures on amplitude integrated electroencephalography
* Exclusion Criteria:

  * A congenital and the hereditary disease, a chromosome abnormalities, and a congenital abnormality.
  * During the acute phases of intracranial and (or) fundus hemorrhage. o
  * Intracranial infection.
  * Pneumothorax.
  * Infants who have been received hypothermia.

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Number of Death or Moderate to Severe Disability Which is Graded According to Gross Motor Function Classification System （GMFCS） | 18 months of life
  Number of Death or Moderate to Severe Disability Which is Graded According to

SECONDARY OUTCOMES:
Number of Infants with abnormal ambulatory electroencephalography monitoring Abnormalities | 3 months of life
  Number of Infants with abnormal ambulatory electroencephalography monitoring
Number of Infants with Brain Magnetic Resonance Imaging Abnormalities | 3 months of Lif
  Number of Infants with Brain Magnetic Resonance Imaging Abnormalities
Number of Infants with Brain-stem Auditory Evoked Potentials Abnormalities at 3 Months of Life | 3 months of life
  Number of Infants with Brain-stem Auditory Evoked Potentials
neonatal behavioral neurological assessment | 7,14 and 28 days after birth
  neonatal behavioral neurological assessment
Bayley Scales of Infant Development | 6,12 and 18 months of life
  Bayley Scales of Infant Development
Gross Motor Function Classification System | 18 months of life
  Gross Motor Function Classification System
Adverse Events That Are Related to Treatment | 3 months of life
  fundus examination by ophthalmofunduscope to evaluate retinopathy of prematurity，chest radiograph to evaluate pneumothorax, and monitoring vital signs by neonatal monitor

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Huang, Doctor, Study Chair — Nanfang Hospital, Southern Medical University
Locations (10):
- China (10):
  - Xiamen Maternity and Child Healthcare Hospital, Xiamen, Fujian
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Maternity and Child Healthcare Hospital, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The Maternity and Child Healthcare Hospital of Guangxi Zhuang Autonomous Region, Guangxi, Guangxi
  - Hunan Children's hospital, Changsha, Hunan
  - The First Hospital of Jilin University, Jilin, Jilin
  - Chengdu Women and Children's central hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No